CLINICAL TRIAL: NCT05351892
Title: A Combined Single- and Multiple-dose, Open-label, Randomized, 2 x 2 Crossover Study to Investigate the Relative Bioavailability, the Safety and the Tolerability of Elinzanetant (BAY 3427080) in Healthy Female and Male Participants
Brief Title: A Study to Learn More About How Much of the Study Treatment Elinzanetant (or BAY3427080) Gets Absorbed, How Safe it is and How it Affects the Body in Healthy Female and Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22050
Record Dates: First submitted 2022-04-25; First posted 2022-04-28 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men; Hot Flashes; Healthy Volunteers
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A-B (Experimental): Participants will receive a single dose of elinzanetant supplied in strength level 1 and 9 subsequent multiple doses from Days 4 to 12 of Period 1; followed by a single dose of elinzanetant supplied in strength level 2 and 9 subsequent multiple doses from Days 4 to 12 of Period 2.
  Interventions: Drug: Elinzanetant (BAY3427080)
- Treatment B-A (Experimental): Participants will receive a single dose of elinzanetant supplied in strength level 2 and 9 subsequent multiple doses from Days 4 to 12 of Period 1; followed by a single dose of elinzanetant supplied in strength level 1 and 9 subsequent multiple doses from Days 4 to 12 of Period 2.
  Interventions: Drug: Elinzanetant (BAY3427080)

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Soft gel capsule, oral

SUMMARY:
Researchers are looking for a better way to treat men and women with vasomotor symptoms, a condition of having hot flashes caused by hormonal changes.

The study treatment, elinzanetant, is under development to treat symptoms caused by hormonal changes. It works by blocking a substance called neurokinin from sending signals to other parts of the body, which is thought to play a role in starting hot flashes.

Participants of this study will be healthy and will have no benefit from administration of elinzanetant. This study, however, will provide information on how to use elinzanetant in people with vasomotor symptoms.

In previous studies, capsules containing smaller amounts of elinzanetant have been used. To reach the daily dose intended for treatment, 3 of these capsules had to be taken once a day. To reduce the pill burden and make it easier for patients to stick to the treatment, capsules with a higher amount of elinzanetant have been developed.

The main purpose of this study is to learn how much of the study treatment elinzanetant gets into the participants' blood when the same dose is taken as new capsule formulation compared to the old capsule formulation.

To answer this question, the researchers will compare:

* The (average) total level of elinzanetant in the blood (also called AUC)
* The (average) highest level of elinzanetant in the blood (also called Cmax) between both capsule formulations after taking one dose of each.

In addition, the researchers want to compare how much of the new and old elinzanetant formulations get into the blood after intake for 9 subsequent days.

All participants will take both formulations by mouth during the study. Each participant will be in the study for up to 12 weeks, including 10 treatment days for each formulation. Participants will stay in-house for 14 days per capsule formulation. In addition, one screening visit to the study site is planned.

During the study, the study doctor and their team will:

* Do physical examinations
* Take blood and urine samples
* Check vital signs
* Examine the participants' heart health using electrocardiogram (ECG)
* Ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. The study doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 45 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation of the investigator, including medical history, physical examination, blood pressure, pulse rate, body temperature, laboratory tests, and cardiac monitoring
* Body weight of at least 50 kg and body mass index (BMI) within the range 18 to 30 kg/m^2 (inclusive)
* Male or female
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention(s) will not be normal
* Known or suspected allergy or hypersensitivity to elinzanetant or any of their excipients
* Any history of or ongoing endocrine disease
* Any known impairment of testosterone synthesis and metabolism
* Poor venous access
* History of alcohol or drug abuse
* Regular use of prescription drugs, over-the-counter drugs, supplements (e.g. carnitine products, anabolics, high dose vitamins) or herbal products within 2 weeks or 5 half-lives (whichever longer) prior to the first study intervention administration
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them within 4 weeks prior to the first study intervention administration, e.g. any investigational drug, any CYP3A4 inducers including St John's Wort, any proton pump inhibitors, or any other drug known to induce liver enzymes (e.g. dexamethasone, barbiturates), and 2 weeks for any drug known to inhibit liver enzymes (e.g. itraconazole, macrolides) as well as grapefruit.
* Clinically relevant findings in the Electrocardiogram (ECG), such as second or third degree AV block, prolongation of ECG parameters (QTcF > 450 msec, QRS > 120 msec)
* Clinically relevant deviations of the screened laboratory parameters from reference ranges at screening or Day -1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from zero to infinity of elinzanetant after single dose administration (AUC) | 0 to 84 hours after first dose on Study Day 1
  AUC from time 0 to the last data point greater than lower limit of quantification (LLOQ) (AUC[0-tlast]) will be used as a primary parameter, if AUC cannot be determined in all participants.
Maximum observed drug concentration of elinzanetant in plasma after single dose administration (Cmax) | 0 to 84 hours after first dose on Study Day 1

SECONDARY OUTCOMES:
Area under the concentration versus time curve from administration of last dose until 24 hours after last dose of multiple dosing (AUC[0-24]md) | 0 to 24 hours post-dose on Study Day 12/13
Maximum observed drug concentration of elinzanetant in plasma after multiple dose administration (Cmax,md) | 0 to 24 hours post-dose on Study Day 12/13
Observed drug concentration of elinzanetant in plasma prior to next dose administration (Ctrough) | 0 to 24 hours post-dose on Study Day 12/13
Number of participants with treatment-emergent adverse events (TEAEs) | After first administration of study intervention until follow up (Day 14 of Period 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.